CLINICAL TRIAL: NCT02513212
Title: A Clinical Study to Determine the Safety and Effectiveness of Dentinal Hypersensitivity Treatment With Two Different Toothbrushes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015059
Record Dates: First submitted 2015-07-30; First posted 2015-07-31 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Dentin Sensitivity
Keywords: Sensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- oxalate liquid, SnF2 paste, manual toothbrush (Other): Potassium oxalate liquid, professionally applied Stannous fluoride paste, self applied Manual toothbrush
  Interventions: Device: Potassium Oxalate; Drug: Stannous fluoride paste; Device: Manual toothbrush
- oxalate liquid, SnF2 paste, power toothbrush (Other): Potassium oxalate liquid, professionally applied Stannous fluoride paste, self applied Power toothbrush
  Interventions: Device: Potassium Oxalate; Drug: Stannous fluoride paste; Device: Power toothbrush

INTERVENTIONS:
Device: Potassium Oxalate — Professionally applied liquid
Drug: Stannous fluoride paste — SnF2 Paste
Device: Manual toothbrush — Marketed manual toothbrush
  Arms: oxalate liquid, SnF2 paste, manual toothbrush
Device: Power toothbrush — Marketed power toothbrush
  Arms: oxalate liquid, SnF2 paste, power toothbrush

SUMMARY:
This study will determine the effects toothbrush type (power or manual) has on the safety and effectiveness of professional dentinal hypersensitivity treatment with a marketed oxalate-containing solution.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age;
* provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* complete a photography consent agreement pertaining to the collection and use of non-identifying intraoral photographs;
* be in good general health as determined by the Investigator/designee; and
* have at least one tooth with a Schiff sensitivity score of at least 1 in response to the cool air challenge.

Exclusion Criteria:

* self-reported pregnancy or nursing;
* severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* active treatment of periodontitis;
* any diseases or conditions that might interfere with the safe completion of the study; or
* an inability to undergo any study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chad J Anderson DMD Inc, Fresno, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxalate Liquid, SnF2 Paste, Manual Toothbrush | Oxalate Liquid, SnF2 Paste, Power Toothbrush
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxalate Liquid, SnF2 Paste, Manual Toothbrush | Oxalate Liquid, SnF2 Paste, Power Toothbrush | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (14.74) | 46.7 (9.63) | 44.6 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 7 | 8 | 15
  Ethnicity: Black | 1 | 0 | 1
  Ethnicity: Asian Oriental | 2 | 1 | 3
  Ethnicity: Multi-Racial | 1 | 1 | 2
  Ethnicity: Hispanic | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Air Challenge
Description: The Schiff Sensitivity Scale was assessed for each test tooth via an evaporative air challenge. The examiner recorded the Schiff Index score corresponding to the response to the air challenge. The Schiff Index Sensitivity scale is scored as follows- 0: tooth/subject did not respond to stimulus, 1: tooth/subject responds to stimulus, but does not request discontinuation of stimulus, 2: tooth/subject responds to stimulus and requests discontinuation or moves form stimulus, 3: tooth/subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus. The higher the Schiff score, the more sensitive the tooth. The mean change from Baseline was calculated for this measure.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxalate Liquid, SnF2 Paste, Manual Toothbrush | Oxalate Liquid, SnF2 Paste, Power Toothbrush
Number analyzed (Participants) | 11 | 12
Units on a scale | -0.409 (0.701) | -0.917 (0.733)

2. Secondary Outcome: Change From Baseline Visual Analog Scale
Description: Visual Analog Scale (VAS) - subjects are asked to look at a VAS and designate the level of hypersensitivity they experienced as a result of the thermal and water challenges using a continuum scale of 0 = No tooth pain up to 100 = Worst tooth pain ever experienced.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Oxalate Liquid, SnF2 Paste, Manual Toothbrush | Oxalate Liquid, SnF2 Paste, Power Toothbrush
Number analyzed (Participants) | 11 | 12
Units on a scale | -11.000 (12.929) | -28.500 (21.075)

ADVERSE EVENTS:
Arm/Group | Oxalate Liquid, SnF2 Paste, Manual Toothbrush | Oxalate Liquid, SnF2 Paste, Power Toothbrush
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes